CLINICAL TRIAL: NCT02387307
Title: A Phase I Open-Label, Non-Randomized, Dose-Escalation Study of rSIFN-co in Subjects With Advanced Solid Tumors and With an Expansion Cohort at Recommended Dose (RD) in Subjects With Non-Small Cell Lung Cancer, Renal Cell Carcinoma, Melanoma, Hepatocellular Carcinoma or Colon Cancer
Brief Title: A Study of rSIFN-co in Subjects With Advanced Solid Tumors
Acronym: rSIFN-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Huiyang Life Science and Technology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rSIFN-01
Record Dates: First submitted 2015-02-06; First posted 2015-03-13 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Melanoma; Carcinoma, Hepatocellular; Colon Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Melanoma; Carcinoma, Hepatocellular; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort: Dose-Escalation and Expansion (Experimental): Dose-Escalation: Dose escalation in solid tumors utilizing a "3+3" design with intra-subject dose escalation. 4 dose levels of rSIFN-co are planned for determining the RD. Dose of rSIFN-co: 15, 21, 24, 27 and 30 ug.
  Dose-Expansion: The Expansion Cohort will be initiated at the RD. Depending on the RD, the lead in period will occur accordingly. After the lead in period, a period from Cycle 1 to the final administration will be performed as the Treatment Phase during which subjects will undergo a standardized evaluation for the safety and efficacy of rSIFN-co at the RD. Follow-up evaluations will be performed 28 days (±5 days) after the last rSIFN-co administration.
  Interventions: Drug: rSIFN-co

INTERVENTIONS:
Drug: rSIFN-co — rSIFN-co is a drug developed by Sichuan Huiyang Life Science and Technology Corporation for the treatment of solid tumors especially in non-small cell lung cancer and other tumor types. The study comprises of 2 stages: the dose-escalation stage and dose expansion stage.
  Other Names: Recombinant-Compound Interferon (rSIFN-co)

SUMMARY:
This is a multicenter, open-label, phase I study of rSIFN-co (3 times a week via subcutaneous injection for 21 days, with 1 week of washout per cycle).

DETAILED DESCRIPTION:
The Dose-Escalation Cohort will consist of the Pretreatment Phase, the Treatment Phase, the Extension Phase, Discontinuation and Follow-up. The Pretreatment Phase will include a Consent and Screening Period. The Treatment Phase will consist of the Lead in Period and first 21-day cycle of treatment during which subjects will be monitored for the development of dose-limiting toxicity (DLT) following 1 week of washout. The Extension Phase will start from the start of Cycle 2 with intra-subject dose-escalation performed until discontinuation of study treatment. Upon discontinuation of study treatment, discontinuation visit assessments should occur within 7 days of treatment discontinuation or confirmation of discontinuation criteria. End of treatment information will also be collected for all subjects who discontinue treatment after completion of cycle 1 treatment. Follow-up visit/final visit evaluations will be performed 28 (±5 days) days after the last rSIFN-co administration. The decision to undergo dose-escalation to the next dose level will be based on the safety information obtained during Cycle 1.

Dose escalation in solid tumors utilizing a "3+3" design with intra-subject dose escalation. 4 dose levels of rSIFN-co are planned for determining the RD. 3-6 subjects will be assigned to each dose level and followed up for 4 weeks after starting administration in Cycle 1. Each cohort will be started after the tolerability of that dose level has been confirmed in subjects with advanced solid tumors. For subjects starting in the lower dose cohorts, intra-subject dose escalation will be allowed till grade 3/4 toxicity is encountered or highest dose level (after safety and tolerability are confirmed) TIW is reached. In order to minimize the risk of allergic reactions, the sponsor has advised a lead-in period starting from 15μg. When the tolerability of each dose level has been confirmed by the observation of no DLT among 3 subjects, escalation to the next dose level will occur.

The Expansion Cohort will be initiated at the RD. Depending on the RD, the lead in period will occur accordingly. After the lead in period, a period from Cycle 1 to the final administration will be performed as the Treatment Phase during which subjects will undergo a standardized evaluation for the safety and efficacy of rSIFN-co at the RD. If subjects are discontinued from the study treatment, discontinuation visit assessments should occur within 7 days of last rSIFN-co administration or confirmation of discontinuation criteria. End of treatment information will also be collected for all subjects who discontinue treatment after completion of cycle 1 treatment. Follow-up evaluations will be performed 28 days (±5 days) after the last rSIFN-co administration.

ELIGIBILITY:
Inclusion Criteria:

1. a) Histologically confirmed diagnosis of advanced solid tumors that is metastatic or unresectable and for which standard therapies (according to local practice) or palliative measures do not exist or subject decides not to receive any available treatment (dose escalation cohort) OR

   b) Histologically or Cytologically diagnosis of Non-Small Cell Lung Cancer, Renal Cell Carcinoma, Melanoma, Hepatocellular Carcinoma* and Colon Cancer metastatic or unrespectable and for which standard therapies (according to local practice) or palliative measures do not exist or subject decides not to receive any available treatment (dose expansion cohort) (dose expansion cohort)

   * Hepatocellular Carcinoma patients may be enrolled based on radiological diagnosis instead of histological or cytological diagnosis - based on "EASL-EORTC Clinical Practice Guidelines: Management of hepatocellular carcinoma (Journal of Hepatology 56:908-943, 2012), non-invasive hepatocellular carcinoma patients should not be put under additional undue risk of liver biopsy after the diagnosis of hepatocellular carcinoma has been ascertained with clinical, laboratory and radiographic evaluation."
2. Measurable disease is preferred but not mandatory for the purpose of study accrual. Evaluable disease is sufficient.
3. Age > or = 21 years
4. ECOG performance status < or = 2
5. Adequate laboratory values at the time of screening:

   (For both dose escalation and expansion)
   * leukocytes ≥3,000/mcL
   * absolute neutrophil count ≥1,500/mcL
   * platelets ≥100,000/mcL
   * haemoglobin ≥9.0 g/DL

   (Dose escalation only)
   * total bilirubin ≤ the upper limits of normal (ULN)
   * AST(SGOT)/ALT(SGPT) ≤ the upper limits of normal (ULN)
   * creatinine < the upper limits of normal (ULN) OR creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal

   (Dose expansion only)
   * total bilirubin ≤ 1.5 times the upper limits of normal (ULN)
   * AST(SGOT)/ALT(SGPT) ≤ 2.5 times the upper limits of normal (ULN) or ≤ 4 times upper limits of normal (ULN) for patients with liver metastasis
   * creatinine ≤1.5 times the upper limits of normal (ULN) OR creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above 1.5 times the institutional upper limits of normal

   (For renal cell carcinoma patients)
   * creatinine ≤ 1.5 times the upper limits of normal (ULN) OR creatinine clearance ≥ 40 mL/min/1.73 m2 for subjects with creatinine levels above 1.5 times the institutional upper limits of normal.
6. Life expectancy > 3 months
7. Agreement to be compliant to visit schedules as defined in the protocol.
8. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.
9. The effects of rSIFN-co on the developing human fetus are unknown. For this reason women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of r-SIFN-co administration. WOCBP must have a negative urine pregnancy test at Visit 1 (Screening).

Exclusion Criteria:

1. Subjects who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to start of rSIFN-co administration or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Subjects receiving other investigational drugs within 5 times the half-life of the investigational drugs or within 4 weeks, prior to start of rSIFN-co administration.
3. Subject must not have known untreated brain or meningeal metastases. CT scans are not required to rule out brain or meningeal metastases unless there is a clinical suspicion of central nervous system disease. Subjects with treated brain metastases that are radiographically or clinically stable for at least 4 weeks after therapy and have no evidence of cavitation or hemorrhage in the brain lesion(s) are eligible, provided that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 4 weeks prior to start of rSIFN-co administration).
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to interferon.
5. Uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, interstitial pneumonia or psychiatric illness/social situations that would limit compliance with study requirements.
6. HIV-positive subjects on combination antiretroviral therapy are ineligible because of the increased risk of lethal infections when treated with immunomodulatory therapy. Appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated.
7. The investigator or sub-investigator considers the subject's physique as inappropriate for investigational product treatment or any other reason(s) that may render the subjects inappropriate for participation in the trial.
8. Subjects who may have autoimmune disorders, decompensated liver diseases or life-threatening neurologic diseases.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events of rSIFN-co of recombinant interferon-α administered in solid Tumor | Up to 12 weeks after the last treatment
  Safety and tolerability will be determined after each cycle of treatment with SIFN-co of recombinant interferon-α, to patients via subcutaneous injection for 21 days (up to 6 cycles)
Recommended dose (RD) of rSIFN-co | Cycle 1 of treatment
  3+3 design for determination of RD. 4 doses (21µg, 24µg, 27µg and 30µg) are planned for determination of RD, dose escalation will be allowed till grade 3/4 toxicity is encountered in 2 or more of the 3 or 6 subjects in first cycle of treatment cycle

SECONDARY OUTCOMES:
Antitumor efficacy (Disease Control Rate), i.e. the percentage of patients, on the RD of rSIFN-co | Up to 28 days after the last treatment
  Antitumor response will be evaluated based on RECIST and irRC guidelines
Objective response rate (ORR), i.e. the percentage of patients, on rSIFN-co | Up to 28 days after the last treatment
  Subjects will be re-evaluated at end of cycle 1, completion of every even cycle treatment, Discontinuation Visit and Follow-up Visit. Confirmatory scans will be obtained within 4 to 8 weeks following initial documentation of an objective response. Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009].
  Antitumor response based on total measurable tumor burden irRC, index and measurable new lesions are taken into account. Each subsequent tumor assessment, the SPD of the index lesions and of new, measurable lesions (≥5 × 5 mm; up to 5 new lesions per organ: 5 new cutaneous lesions and 10 visceral lesions) are added together to provide the total tumor burden, the objective is to determine response rate (ORR), progression-free survival (PFS),and time to progression (TTP) status on rSIFN-co.
Progression-free survival (PFS) time (days) on rSIFN-co | Up to 28 days after the last treatment
  Subjects will be re-evaluated at end of cycle 1, completion of every even cycle treatment, Discontinuation Visit and Follow-up Visit. Confirmatory scans will be obtained within 4 to 8 weeks following initial documentation of an objective response. Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009].
  Antitumor response based on total measurable tumor burden irRC, index and measurable new lesions are taken into account. Each subsequent tumor assessment, the SPD of the index lesions and of new, measurable lesions (≥5 × 5 mm; up to 5 new lesions per organ: 5 new cutaneous lesions and 10 visceral lesions) are added together to provide the total tumor burden, the objective is to determine response rate (ORR), progression-free survival (PFS),and time to progression (TTP) status on rSIFN-co.
Time to progression (TTP) status (days) on rSIFN-co | Up to 28 days after the last treatment
  Subjects will be re-evaluated at end of cycle 1, completion of every even cycle treatment, Discontinuation Visit and Follow-up Visit. Confirmatory scans will be obtained within 4 to 8 weeks following initial documentation of an objective response. Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009].
  Antitumor response based on total measurable tumor burden irRC, index and measurable new lesions are taken into account. Each subsequent tumor assessment, the SPD of the index lesions and of new, measurable lesions (≥5 × 5 mm; up to 5 new lesions per organ: 5 new cutaneous lesions and 10 visceral lesions) are added together to provide the total tumor burden, the objective is to determine response rate (ORR), progression-free survival (PFS),and time to progression (TTP) status on rSIFN-co.
FDG-PET response (lesion size) before and after administration of rSIFN-co | Up to 28 days after the last treatment
  CT and SUV values used to determine lesion size will be evaluated and studied to understand the change of CT value& SUV value before and after treatment.
FDG-PET response (lesion volume) before and after administration of rSIFN-co | Up to 28 days after the last treatment
  CT and SUV values used to determine lesion volume will be evaluated and studied to understand the change of CT value& SUV value before and after treatment.

OTHER OUTCOMES:
Changes in subject cytokine profiles (pg/ml) before and after treatment | Up to 28 days after the last treatment
  The cytokine data is an experimental observation and not used for therapeutic effect evaluation. if possible, to evaluate the correlation between these cytokine changes and study drugs.
Evaluation of elected tumor repressive and enhancing genes (counts of genes such as microRNA-92a, microRNA-92b) before and after administration of rSIFN-co | Up to 28 days after the last treatment
  Pre- and post-dose samples will be collected for additional cell signaling assays to evaluate selected tumor repressive and enhancing genes (such as microRNA-92a, microRNA-92b) as well as levels of 2'5'-oligoadenylate synthetase.
Evaluation of levels (counts) of 2'5'-oligoadenylate synthetase, before and after administration of rSIFN-co | Up to 28 days after the last treatment
  Pre- and post-dose samples will be collected for additional cell signaling assays to evaluate selected tumor repressive and enhancing genes (such as microRNA-92a, microRNA-92b) as well as levels of 2'5'-oligoadenylate synthetase.

CONTACTS AND LOCATIONS:
Overall Officials: David Wai Meng TAI, Principal Investigator — National Cancer Center Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided